CLINICAL TRIAL: NCT02140203
Title: Effect of Yoga on Metabolic Abnormalities Outcomes in Middle-Aged and Older Adults With Metabolic Syndrome
Brief Title: Effects of Yoga on Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Angus Yu (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Sponsor-Investigator, Angus Yu, Project Assistant, The Hong Kong Polytechnic University
Organization: The Hong Kong Polytechnic University (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: MetsYoga
Record Dates: First submitted 2014-05-13; First posted 2014-05-16 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome; Waist circumference; blood pressure; triglyceride; HDL
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Young Yoga Group (Active Comparator): People who are younger than 60 year-old They have received Yoga training in one-year experimental period
  Interventions: Other: Yoga Training
- Young Control Group (No Intervention): People who are younger than 60 year-old No Yoga training through out the one-year experimental period
- Aged Control Group (No Intervention): People who are equal or older than 60 year-old They have not received any yoga training during the one-year experimental period
- Aged Yoga Group (Active Comparator): People who are equal or older than 60 year-old They have received any yoga training during the one-year experimental period
  Interventions: Other: Yoga Training

INTERVENTIONS:
Other: Yoga Training — one-year experimental training (three times per week and one hour per session)
  Other Names: Hatha Yoga Training
  Arms: Aged Yoga Group; Young Yoga Group

SUMMARY:
Metabolic syndrome (MetS) is a clustering of cardiovascular risk factors characterizing central obesity, insulin resistance, dyslipidemia and high blood pressure. The concept of MetS represents the pre-cardiovascular and pre-diabetic pathologic conditions, which has been a useful tool in prognosing the development of cardiovascular disease and diabetes mellitus. Importantly, interventions applied at the pre-pathologic stage with MetS would be of great clinical and health significance in achieving better preventive and therapeutic outcomes. Yoga, a mind-body exercise, has been suggested to have beneficial effects on dyslipidemia, hypertension and diabetes. A pilot study has demonstrated the trends in the improvement of metabolic parameters in middle-aged adults with MetS but the findings are inconclusive because of the small sample size and brief yoga follow-up period (i.e., 2-month). In addition to the needs of a better designed randomized controlled trial in studying the beneficial effect of yoga in controlling MetS in middle-aged individuals, the investigation on yoga and MetS in elderly population has been lacking. This is important as the potential use of yoga as lifestyle modification in elderly individuals with MetS will result in significant reduction of the prevalence of cardiovascular disease and diabetes. Thus, this study aims to examine the efficacy of yoga exercise in improving metabolic abnormalities in middle-aged and older adults with MetS. In addition to elderly, middle-aged adults are included in the present investigation because of the idea that cardiovascular diseases and diabetes with aging can be mostly prevented by intervention at the middle-age. A randomized controlled trial with repeated measure design will be conducted to examine the effect of 1-year regular yoga training on the MetS parameters in middle-aged and older individuals who are 30-60 and 60-80 years of age, respectively. Primary outcome measures include waist circumference, systolic/diastolic blood pressure, blood glucose, triglyceride, and lipid cholesterol profile whereas secondary outcome measures include self-reported stress and depression levels. This study is anticipated to provide valuable information in exploring the therapeutic role of yoga in managing MetS. As yoga exercise is an economical regimen which can be easily and readily applied to large scale of target population, it is of hope to be practically useful to relieve the burden on cardiovascular disease and diabetes by introducing yoga lifestyle to the management of MetS.

ELIGIBILITY:
Inclusion Criteria:

MetS is defined as having three or more (>= 3) of the following conditions:

* Central obesity - Waist circumference >= 90 cm (Asian male); 80 cm (Asian female)
* High blood pressure - Systolic blood pressure/diastolic blood pressure >= 130/85 mmHg or use of hypertension drug
* Elevated blood glucose - Fasting blood glucose >= 100 mg/dL or use of hyperglycemia drug
* Elevated blood triglyceride - Blood triglyceride >= 150 mg/dL
* Reduced HDL-cholesterol - HDL-C <= 40 mg/dL (male); <= 50 mg/dL (female)

Exclusion Criteria:

* Dementia
* Mental disorders
* Severe or acute cardiovascular illnesses
* Post-stroke,
* Neuromusculoskeletal illnesses
* Major orthopaedic diagnosis in the lower back
* Pelvis or lower extremities
* Severe rheumatoid arthritis
* Osteoarthritis
* Pulmonary illnesses
* Immobile
* Wheelchair users
* Undertaking drug therapy treating metabolic abnormalities
* Acute medical illness
* Symptomatic heart disease
* Symptomatic lung disease
* Physical conditions not suitable for exercise training, and tobacco users
* Regular physical activities (>= 3 days per week of moderate exercise intensity >= 30 minutes)

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2010-07; Primary Completion 2011-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in waist circumference | Six Months
  The operational definition of waist circumference is the measure of circumference at the waist area. This is a commonly used indicator for recognizing central obesity. The waist circumference will be determined by using tape with metric scale. To determine the waist circumference, the upper hip bone will be located and a measuring tape will be placed around the abdomen. The tape measure will be horizontal and the measuring tape will not be snug but without causing compressions on the skin.
Change in systolic/diastolic blood pressure | Six Months
  Resting blood pressure measurement will be performed after the subject has taken 15-minute rest in the laboratory by using an electronic blood pressure monitor. Both the systolic and diastolic blood pressure will be obtained with the cuff over brachial artery region at the level of heart.
Change in blood glucose | Six Months
  Measurements will be performed on the glucose and insulin level in venous blood sample collected after overnight fast. Subjects will be asked to come to the laboratory after an overnight ~10 hours fasting. Before each resting blood sampling, subjects will be requested to sit in a quiet environment for 15 minutes prior to blood collection. Ten ml of venous blood will be drawn from an antecubital vein in the forearm. The blood collection will be performed by a licensed nurse or medical lab technologist. After collection of venous blood sample, blood samples will be dispensed into a lithium heparin plastic tube to prevent coagulation. The remnant whole blood will be centrifuged to obtain plasma samples and stored at -80°C in a freezer before being analyzed for glucose
Change in triglyceride | Six Months
  Ten ml of venous blood will be drawn from an antecubital vein in the forearm. The blood collection will be performed by a licensed nurse or medical lab technologist. After collection of venous blood sample, blood samples will be dispensed into a lithium heparin plastic tube to prevent coagulation. The remnant whole blood will be centrifuged to obtain plasma samples and stored at -80°C in a freezer before being analyzed for triglyceride.
Change in lipoprotein | Six Months
  The blood collection will be performed by a licensed nurse or medical lab technologist. After collection of venous blood sample, blood samples will be dispensed into a lithium heparin plastic tube to prevent coagulation. Measurements will be performed on HDL-C level in the collected venous blood samples.
Change in waist circumference | One year
  The operational definition of waist circumference is the measure of circumference at the waist area. This is a commonly used indicator for recognizing central obesity. The waist circumference will be determined by using tape with metric scale. To determine the waist circumference, the upper hip bone will be located and a measuring tape will be placed around the abdomen. The tape measure will be horizontal and the measuring tape will not be snug but without causing compressions on the skin.
Change in systolic/diastolic pressure | One year
  Resting blood pressure measurement will be performed after the subject has taken 15-minute rest in the laboratory by using an electronic blood pressure monitor. Both the systolic and diastolic blood pressure will be obtained with the cuff over brachial artery region at the level of heart.
Change in blood glucose | One year
  Measurements will be performed on the glucose and insulin level in venous blood sample collected after overnight fast. Subjects will be asked to come to the laboratory after an overnight ~10 hours fasting. Before each resting blood sampling, subjects will be requested to sit in a quiet environment for 15 minutes prior to blood collection. Ten ml of venous blood will be drawn from an antecubital vein in the forearm. The blood collection will be performed by a licensed nurse or medical lab technologist. After collection of venous blood sample, blood samples will be dispensed into a lithium heparin plastic tube to prevent coagulation. The remnant whole blood will be centrifuged to obtain plasma samples and stored at -80°C in a freezer before being analyzed for glucose
Change in triglyceride | One year
  Ten ml of venous blood will be drawn from an antecubital vein in the forearm. The blood collection will be performed by a licensed nurse or medical lab technologist. After collection of venous blood sample, blood samples will be dispensed into a lithium heparin plastic tube to prevent coagulation. The remnant whole blood will be centrifuged to obtain plasma samples and stored at -80°C in a freezer before being analyzed for triglyceride.
Change in lipoprotein | One year
  The blood collection will be performed by a licensed nurse or medical lab technologist. After collection of venous blood sample, blood samples will be dispensed into a lithium heparin plastic tube to prevent coagulation. Measurements will be performed on HDL-C level in the collected venous blood samples.

SECONDARY OUTCOMES:
Change in self-reported stress and depression levels | Six Months
  Self-reported stress and depression levels are proposed to be the secondary outcome measures because the stress and depression levels could be improved by yoga intervention which might have beneficial effects on MetS parameters indirectly. The indicator of stress level will be adopted to estimate the mental health in this project. The Patton Type A personality questionnaire will be used to examine the stress level. The Center for Epidemiologic Studies Depression Scale (CES-D) will be used to estimate the depression level of the subjects.
Change in Self-reported stress and depression levels | One year
  Self-reported stress and depression levels are proposed to be the secondary outcome measures because the stress and depression levels could be improved by yoga intervention which might have beneficial effects on MetS parameters indirectly. The indicator of stress level will be adopted to estimate the mental health in this project. The Patton Type A personality questionnaire will be used to examine the stress level. The Center for Epidemiologic Studies Depression Scale (CES-D) will be used to estimate the depression level of the subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Parco MF Siu, PHD, Principal Investigator — Associate Professor, Department of Health Technology and Informatics, The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, China